CLINICAL TRIAL: NCT01871610
Title: Amyloid Accumulation After Mild Traumatic Brain Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 100-4313A
Record Dates: First submitted 2013-05-02; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; mild TBI; Alzheimer's disease; [18F]AV-45 PET amyloid binding imaging
MeSH Terms: conditions — Brain Injuries, Traumatic; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alzheimer disease after mild traumatic brain injury (Experimental): Based on the TBI registry databank, to recruit patients 1, 5, 10, 15 years after mTBI for cognitive evaluatio
  Interventions: Drug: [18F]AV-45 PET amyloid binding imaging
- mild traumatic brain injury without Alzheimer disease (Experimental): To recruit patients 1, 5, 10, 15 years after mTBI with or without cognitive impairment and age-gender-matched controls (a total of 3 groups) for amyloid- positron emission tomography (A-PET)
  Interventions: Drug: [18F]AV-45 PET amyloid binding imaging
- Normal control (Experimental): People aged 30 or older without mTBI or AD
  Interventions: Drug: [18F]AV-45 PET amyloid binding imaging

INTERVENTIONS:
Drug: [18F]AV-45 PET amyloid binding imaging

SUMMARY:
There will be 200 participants, who aged 30 years or older with TBI in 1,5,10,15 years ago and GCS=13-15 will be recruited. Another group of 200 participants with the same age and gender and without TBI will be recruited as the controls. All of them will undergo AD8 questionnaire for dementia screening and APOE4 genotyping. Further CASI and CDR will be tested for the confirmation of dementia diagnosis for the individuals with AD8 scaore >/=2. 10 TBI with dementia, 20 TBI without dementia and 10 controls will be selected randomly for AV45 amylid PET study.

There will also be 10 participants without traumatic brain injury and interested in this study, aged 55 years or older better.

DETAILED DESCRIPTION:
We will examine the mTBI patients in a long-term follow-up manner by cognitive tests and A-PET. This is a novel study for linking mTBI and AD by solid, reliable methods, in terms of A-PET and cognitive function tests. In addition, we will figure out the importance of APOE genotypes for amyloid accumulation and cognitive impairment. These results should shed light on the further clinical studies and amyloid-cleaning therapy for prevention and treatment for dementia after mTBI.

ELIGIBILITY:
Inclusion criteria:

* The individuals are listed in the Taipei medical university traumatic brain injury databank and had TBI in 1, 5, 10 and 15 years ago. There are about 200 individuals undergo telephone interview/invitation, blood test for genotyping and neuropsychological tests. 30 participants will be selected randomly among the 200 individuals.
* mild injury in TBI (initial GCS = 13-15)
* had MRI or CT evaluation after TBI
* aged 30 years or older better
* agreed by principal investigator
* have agreement and have signed the informed consent form by him/herself or his/her legal representative

Main exclusion criteria:

* participating in another clinical trials which might interfere the current finding.
* not sure the timing of TBI
* contaminant the symptoms with injury, skull fracture, intracranial hemorrhage, craniotomy, and death
* moderate (initial GCS = 9-12) or severe (initial GCS < 8) injury in TBI
* had wound with gunshot or puncture
* loss of consciousness over 30 minutes after TBI
* loss of memory for over 1 day after TBI
* have no MRI or CT evaluation of brain after TBI or have obstructive ischemia after MRI or CT evaluation
* have uremia, liver cirrhosis, heart failure, pulmonary edema, coagulation disorders and other major diseases
* pregnant woman or emotional instability
* the age less than 18 years (30 years better)
* unable to collect blood sample by peripheral vein
* determination of inappropriate participants in the clinical trail of PI

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
The amyloids load in brain among mild traumatic brain injury and controls in a temporal manner. | one year
  The amyloids load (based on F-18-AV-45 binding) in brain among mild traumatic brain injury and controls in a temporal manner.

SECONDARY OUTCOMES:
F-18-AV-45 binding changes and cognitive function among mild traumatic brain injury and controls | one year
  To evaluate the the F-18-AV-45 binding in different APOE genotypes among mild traumatic brain injury and controls

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Chen YEN, MD, PhD, Study Director — Nuclear Medicine